CLINICAL TRIAL: NCT00829270
Title: Economic and Medical Evaluation of the Whole Mitochondrial DNA Screening by Surveyor and Mitochips Techniques.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PSTIC Mitochips
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2009-01

CONDITIONS: Mitochondrial Disease
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — patients presenting clinical features of mitochondrial diseases
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mitochondrial diseases diagnosis

SUMMARY:
Mitochondrial diseases are the most frequent metabolic diseases (2.5 persons among 10 000) and are clinically heterogeneous making diagnosis particularly challenging for clinicians.

Molecular analysis of mitochondrial DNA (mtDNA) is a critical step in diagnosis and genetic counselling of respiratory chain defects. DNA sequencing remains the gold standard but it is time-consuming and fails to detect mutations that may be present at a low heteroplasmic level (20% or below); therefore the diagnosis is yet based on the detection of a few number of pathogenic mutations.

The present study aims to evaluate the benefit and the cost of a diagnosis strategy based on the combined use of 2 techniques named "Surveyor Nuclease" and "Mitochip". Surveyor nuclease is a mismatch-specific DNA endonuclease that will be used for screening the entire mtDNA in order to identify heteroplasmic mutations. In absence of any identified mutation, another technique based on the use an oligonucleotide sequencing microarray (MitoChip) will be performed for the identification of homoplasmic mutations. Mitochip is an array-based sequencing platform for rapid and high-throughput analysis of mitochondrial DNA.

The economical study will compare the cost of these techniques to the standard diagnosis method in term of direct and indirect costs

ELIGIBILITY:
Inclusion Criteria:

* patients without deletion of mitochondrial disease and/or 3243, 8344 and 8993 mutation
* patient with health insurance

Exclusion Criteria:

* patients with deletion of mitochondrial disease and/or 3243, 8344 and 8993 mutation
* absence of patient consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting clinical features of mitchondrial diseases
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the benefit and the cost of a mitochondrial disease diagnosis strategy based on the combined use of 2 techniques named "Surveyor Nuclease" and "Mitochip" | 2 years

SECONDARY OUTCOMES:
Evaluation of the benefit of the studiad strategy in comparison with standard diagnosis method in term of indirect costs | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Véronique PAQUIS-FLUCKINGER, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice - Medical genetics laboratory, Nice, France